CLINICAL TRIAL: NCT00355940
Title: Comparing Fluoroscopy and Technological Methods for Guidance During Endovascular Procedures Traditional Fluoroscopy Navigation Based on Preoperative CT and Intraoperative DynaCT
Brief Title: Comparing Fluoroscopy and Technological Methods for Guidance During Endovascular Procedures
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: SINTEF Health Research (Other); St. Olavs Hospital (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STO-NTNU/DMF-SINTEF-1
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: endovascular; aortic; repair; navigation; DynaCT; position; sensor
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Technological Methods
- 2 (Active Comparator)
  Interventions: Device: Regular Fluoroscopy

INTERVENTIONS:
Device: Technological Methods — Usage of technological methods and devices to improve intravascular navigation during endovascular aortic repair.
  In this arm we first use an optical pointer to allocate the femoral artery ramification (point of incision) and the lower renal artery (upper confinement of stent graft). Later we use an electromagnetically tracked catheter to find and enter the opening in the main stent graft before placing the second limb. For both optical and electromagnetic tracking we use a custom made navigation system based on 3 dimensional CT images
  Other Names: Custom made devices in addition to Siemens angiography suite
  Arms: 1
Device: Regular Fluoroscopy — Usage of conventional fluoroscopy and angiography for intravascular navigation. In this arm standard endovascular aortic repair is performed. The only means of navigation are fluoroscopy and angiography with overlay function (standard).
  Other Names: Siemens angiography suite
  Arms: 2

SUMMARY:
The investigators want to test a navigation system for guidance during insertion of stent graft in abdominal aortic aneurysms. The navigation system consists of software developed by SINTEF Health, a custom made catheter with a micro position sensor in the tip and an emitter than induces an electromagnetic field around the patient. Preoperative CT- and intraoperative DynaCT- data are reconstructed into 3 dimensional images. The 3 dimensional images are loaded into the navigation system. Then the magnetic field, in which the patient finds himself, is calibrated with the 3 dimensional images. When the catheter is inserted into the iliac artery and aorta, the position sensor (in the tip of the catheter) is displayed in real time at the exact anatomic location in the 3 dimensional image.

Null hypothesis (H0):

* Insertion of stent graft is performed equally satisfactorily with fluoroscopy alone as with both fluoroscopy and new navigation technology

Alternative hypothesis (H2):

* Insertion of stent graft is NOT performed equally satisfactorily with fluoroscopy alone as with both fluoroscopy and new navigation technology

ELIGIBILITY:
Inclusion Criteria:

* AAA with diameter > 5,0 cm suitable for endovascular technique
* Normal creatinine
* > 60 years of age

Exclusion Criteria:

* Known heart failure or unstable coronary disease
* Other morbidity than normally contraindicates endovascular treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Measure time (s) for defining renal branch | No time frame
Measure time (s) for inserting guidewire into "second limb" | 900 sec
Number of attempts for inserting guidewire into "second limb" | 900 sec
Measure total time (min) for entire procedure | No time frame
Measure the total of x-ray dose (mGy/m2) | No time frame
Measure the total of contrast fluid used (ml) | No time frame
Define type I leak between stent graft and aortic wall | No time frame
Measure distance (mm) between stent graft and renal arteries | No time frame
Measure difference (mm) in actual position and position in 3D image when pointing at the femoral division with an optic pointer | No time frame
Measure difference (mm) of the position of the renal arteries defined by optical pointer and angiography (both marked extracorporal with a needle) | No time frame

SECONDARY OUTCOMES:
1 questionnaire: "Can 3D image and navigation technology simplify and secure endovascular procedures?" | No time frame
2 questionnaire: "Do you believe in further development of this technology?" | No time frame
3 questionnaire: "Have both renal arteries unaltered flow?" | No time frame

CONTACTS AND LOCATIONS:
Overall Officials: Frode Manstad-Hulaas, MD, Principal Investigator — Norwegian University of Science and Technology; Petter Aadahl, Professor, Study Director — Norwegian University of Science and Technology; Toril N Hernes, Professor, Study Director — SINTEF Health Research
Locations (1):
- St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Manstad-Hulaas F, Tangen GA, Dahl T, Hernes TA, Aadahl P. Three-dimensional electromagnetic navigation vs. fluoroscopy for endovascular aneurysm repair: a prospective feasibility study in patients. J Endovasc Ther. 2012 Feb;19(1):70-8. doi: 10.1583/11-3557.1. PMID 22313205